CLINICAL TRIAL: NCT00179348
Title: Evaluation of a Yoga-Based Cancer Rehabilitation Program
Brief Title: Yoga-Based Rehabilitation Program in Reducing Physical and Emotional Side Effects in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000-007; NCI-2014-01579 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000-007; NCI R03 CA88598-01A1; 01-02-038; CCI# 00-7 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH); R03CA088598 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Alopecia; Anxiety; Breast Carcinoma; Cognitive Side Effects of Cancer Therapy; Colorectal Carcinoma; Depression; Fatigue; Lung Carcinoma; Nausea and Vomiting; Pain; Psychological Impact of Cancer; Sleep Disorder; Weight Change
MeSH Terms: conditions — Alopecia; Anxiety Disorders; Breast Neoplasms; Colorectal Neoplasms; Depression; Fatigue; Lung Neoplasms; Nausea; Vomiting; Pain; Sleep Wake Disorders; Body Weight Changes | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (yoga-based rehabilitation program) (Experimental): Participants undergo a yoga-based rehabilitation program up to 5 days a week for 1.5 hours and practice at home at least once daily for 12 weeks.
  Interventions: Procedure: Quality-of-Life Assessment; Procedure: Yoga
- Group II (standard care/control) (Active Comparator): After a 3 month wait period, participants undergo a yoga-based rehabilitation program as in Group I.
  Interventions: Procedure: Quality-of-Life Assessment; Procedure: Yoga

INTERVENTIONS:
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Yoga — Undergo a yoga-based rehabilitation program
  Other Names: Yoga Therapy

SUMMARY:
This clinical trial studies yoga-based rehabilitation in reducing physical and emotional side effects of living with cancer or its treatment. Yoga-based rehabilitation may reduce side effects and improve the quality of life of patients with breast, lung, or colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effects of yoga on quality of life (QOL) of breast cancer patients on different treatment regimens.

II. To pilot the effects of a yoga-based rehabilitation program versus standard care on QOL impairment reported by newly diagnosed (a) lung and (b) colorectal patients.

III. To evaluate program compliance and satisfaction among breast, lung and colorectal cancer patients as well as among the various sociocultural subgroups (e.g., ethnicity, language).

OUTLINE: Participants are randomized to 1 of 2 arms.

GROUP I (YOGA-BASED REHABILITATION PROGRAM): Participants undergo a yoga-based rehabilitation program up to 5 days a week for 1.5 hours and practice at home at least once daily for 12 weeks.

GROUP II (STANDARD CARE/CONTROL): After a 3 month wait period, participants undergo yoga-based rehabilitation program as in Group I.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with breast, lung or colorectal cancer in the previous 8 weeks
* Are to receive oncologic care at the Albert Einstein Cancer Center (AECC)
* Have a life-expectancy of at least 6 months
* Are either English- or Spanish-speaking
* Do not practice yoga regularly (> 1 month)
* Receive medical clearance by oncologic personnel on the study

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status >= 3
* Existence of any of the following:

  * Seizure disorder
  * Musculoskeletal conditions
  * Heart problems
  * Major psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2001-02-08 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy summary score (physical, emotional, spiritual, and social QOL) | Baseline to up to 6 months
  A repeated measures analysis of covariance will be performed for each of the five patient groups. This analysis will examine between and within group differences at T2 and T3 assessment points, after controlling for baseline levels of QOL.
Program compliance as measured by Yoga - Daily Practice Calendar and Yoga Class Attendance Record and Yoga Evaluation Form | Up to 6 months
  Descriptive analyses (percentages) will be conducted to examine levels of compliance (class attendance + home practice) for each patient group, self-identified ethnic group, and language of preference. Logistic regression analyses will be performed to identify patients in the top 25% for compliance based on sociocultural, medical, and lifestyle factors.
Program satisfaction measured by Yoga - Daily Practice Calendar and Yoga Class Attendance Record and Yoga Evaluation Form | Up to 6 months
  Descriptive analyses (percentages) will be conducted to examine levels of satisfaction (total score on yoga evaluation form) for each patient group, self-identified ethnic group, and language of preference. Logistic regression analyses will be performed to identify patients in the top 25% for satisfaction based on sociocultural, medical, and lifestyle factors.

SECONDARY OUTCOMES:
Pain | Baseline to up to 6 months
  Medical chart data will be examined and three separate one-way analysis of variances will be conducted to examine mean differences in adverse medical events, compliance with cancer treatment, and use of pharmacotherapy between intervention and control for each of the five cancer patient groups.
Mood | Baseline to up to 6 months
  Medical chart data will be examined and three separate one-way analysis of variances will be conducted to examine mean differences in adverse medical events, compliance with cancer treatment, and use of pharmacotherapy between intervention and control for each of the five cancer patient groups.
spiritual well-being | Baseline to up to 6 months
  Medical chart data will be examined and three separate one-way analysis of variances will be conducted to examine mean differences in adverse medical events, compliance with cancer treatment, and use of pharmacotherapy between intervention and control for each of the five cancer patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Moadel, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Moadel AB, Shah C, Wylie-Rosett J, Harris MS, Patel SR, Hall CB, Sparano JA. Randomized controlled trial of yoga among a multiethnic sample of breast cancer patients: effects on quality of life. J Clin Oncol. 2007 Oct 1;25(28):4387-95. doi: 10.1200/JCO.2006.06.6027. Epub 2007 Sep 4. PMID 17785709